CLINICAL TRIAL: NCT00702741
Title: A Long-Term Follow-up Study of Chondrogen - Adult Human Stem Cells Delivered by Intra-articular Injection Following Meniscectomy in Subjects 18-60 Years
Brief Title: Follow-up Study of Chondrogen® Delivered by Intra-Articular Injection Following Meniscectomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mesoblast International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 551
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Recovery Following Partial Medial Meniscectomy
Keywords: Knee; Meniscus; Meniscectomy; Mesenchymal Stem Cells; MSCs; Adult Human Stem Cells; Osiris; Chondrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Chondrogen (low dose)
  Interventions: Drug: Chondrogen
- B (Experimental): Chondrogen (high dose)
  Interventions: Drug: Chondrogen
- C (Placebo Comparator): Hyaluronan
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chondrogen — Intra-articular injection of ex vivo cultured adult human mesenchymal stem cells
  Arms: A
Drug: Chondrogen — Intra-articular injection of ex vivo cultured adult human mesenchymal stem cells
  Arms: B
Drug: Placebo — Intra-articular injection of Hyaluronan
  Arms: C

SUMMARY:
The objective of the present study is to establish the long-term safety of an intra-articular injection of human mesenchymal stem cells (hMSCs) (Chondrogen).

DETAILED DESCRIPTION:
The long-term safety of human mesenchymal stem cells (hMSCs) (Chondrogen) has not yet been established. This 3-year follow-up study will provide additional data to gain understanding of the safety of the investigational agent. This study is designed to determine the safety of a single intra-articular injection of 50 million donor-derived hMSCs or 150 million donor-derived hMSCs in suspension with commercial sodium hyaluronan compared to an injection of vehicle (diluted hyaluronan) alone. The injections were performed under the initial study, Protocol No. 550.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have received an injection in Protocol No. 550
* Subject must have completed the 6-month and final 2-year visit in Protocol No. 550
* Subject must provide written informed consent for entry into the extension study
* Subject must provide authorization for use and disclosure of protected health information for entry into the extension study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2008-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Comparison of treatment adverse event rates | Through 3 years

SECONDARY OUTCOMES:
Concomitant Medications | Through 3 years
Visual Analog Scale | Through 3 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - OrthoIndy, Indianapolis, Indiana
  - TRIA Orthopaedic Center, Bloomington, Minnesota
  - Unlimited Research, San Antonio, Texas